CLINICAL TRIAL: NCT05772052
Title: Food Addiction, Binge Eating Disorder and Taste Perception in Subjects With Obesity
Brief Title: Abnormal Eating and Taste Perception in Subjects With Obesity
Acronym: TASTEOB
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 43C002
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: Taste; Obesity; Food addiction; Binge eating; sweet; salty
MeSH Terms: conditions — Obesity; Food Addiction; Bulimia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The identification of safe and effective strategies for weight loss and long-term maintenance is critical to reduce the alarming prevalence of obesity worldwide and mitigate obesity-associated health risks. Specifically, Binge Eating (BE) and Food Addiction (FA) behaviors are well known causes of failed weight loss and weight regain. The definitions of their clinical phenotypes are currently evolving. Recent evidence suggests that food choices, behavior and reward may be driven also by taste perception.

The hypothesis of this study is that subjects with dysfunctional eating behavior have different taste thresholds compared to obese subjects without eating disorders, and that this characteristic influences food choice and eating behavior. Identifying a difference in the taste thresholds between obese with and without eating disorder will allow us to understand why certain individuals over-consume or binge on densely caloric foods and to give them a tailored dietary treatment so as to maintain weight loss for a long time.

The Binge eating and Food Addiction is assessed using Binge Eating Scale and Yale Food Addiction Scale 2.0. Subjects with obesity recruited are divided in 4 groups: without eating disorder, with food addiction (FA), with binge eating (BE) and with FA + BE. In these groups sweet and salty taste will be measured with the 3-Alternative-Forced-Choice method.

ELIGIBILITY:
Inclusion Criteria:

* BMI>30 kg/m2 and <45 kg/m2

Exclusion Criteria:

* uncooperative patients
* heavy smokers
* pregnancy or recent (in the last 6 months) childbirth
* thyroid disorders
* presence of endocrine abnormalities associated with obesity
* current or recent oral, nasal or sinus infections
* major psychiatric disorder even in pharmacological compensation
* patients who had undergone bariatric surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects with obesity referred to Istituto Auxologico Italiano for weight loss program
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
sweet taste recognition threshold | baseline
  The sweet taste recognition threshold is assessed in subjects without eating disorders, with FA,with BE and FA+ BE
salt taste recognition threshold | baseline
  The salt taste recognition threshold is assessed in subjects without eating disorders, with FA,with BE and FA+ BE

SECONDARY OUTCOMES:
prevalence of binge eating (BE) | baseline
  percentage of subjects recruited with BE
prevalence of Food Addiction (FA) | baseline
  percentage of subjects recruited with FA
prevalence of Food Addiction (FA) + Binge Eating (BE) | baseline
  percentage of subjects recruited with FA+BE

CONTACTS AND LOCATIONS:
Overall Officials: Simona Bertoli, MD, Study Chair — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

REFERENCES:
- [Background] Aloi M, Rania M, Rodriguez Munoz RC, Jimenez Murcia S, Fernandez-Aranda F, De Fazio P, Segura-Garcia C. Validation of the Italian version of the Yale Food Addiction Scale 2.0 (I-YFAS 2.0) in a sample of undergraduate students. Eat Weight Disord. 2017 Sep;22(3):527-533. doi: 10.1007/s40519-017-0421-x. Epub 2017 Aug 5. PMID 28780748
- [Background] Arlt JM, Smutzer GS, Chen EY. Taste assessment in normal weight and overweight individuals with co-occurring Binge Eating Disorder. Appetite. 2017 Jun 1;113:239-245. doi: 10.1016/j.appet.2017.02.034. Epub 2017 Feb 24. PMID 28242311
- [Background] Bertoli S, Leone A, Ponissi V, Bedogni G, Beggio V, Strepparava MG, Battezzati A. Prevalence of and risk factors for binge eating behaviour in 6930 adults starting a weight loss or maintenance programme. Public Health Nutr. 2016 Jan;19(1):71-7. doi: 10.1017/S1368980015001068. Epub 2015 May 11. PMID 25958773
- [Background] Proserpio C, Laureati M, Bertoli S, Battezzati A, Pagliarini E. Determinants of Obesity in Italian Adults: The Role of Taste Sensitivity, Food Liking, and Food Neophobia. Chem Senses. 2016 Feb;41(2):169-76. doi: 10.1093/chemse/bjv072. Epub 2015 Dec 15. PMID 26671250